CLINICAL TRIAL: NCT03044288
Title: Evaluation of the Effect of Output on Skin Covered by a New Adhesive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP265_09
Record Dates: First submitted 2017-01-31; First posted 2017-02-07 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 9 (Experimental): This is a sub-study testing the effect of real output applied under two adhesive strips on the skin.
  Standard adhesive strip and a strip with a newly developed adhesive (new adhesive strip)
  Interventions: Other: New adhesive strip; Other: Standard adhesive strip

INTERVENTIONS:
Other: New adhesive strip — This is a strip made of a newly developed adhesive. This adhesive might in the future be part of an ostomy product.
Other: Standard adhesive strip — this is a standard adhesive strip (hydrocolloid). This adhesive is currently used in marketed ostomy devices.

SUMMARY:
The study investigates the impact real output has on peristomal skin covered by a newly developed adhesive and a standard adhesive

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have had an ileostomy for more than one year
4. Have intact skin on the area used in the evaluation
5. Has an ileostomy with a diameter up to (≤) 35 mm
6. Have a peristomal area accessible for application of patches/adhesive strips (assessed by investigating scientist) -

Exclusion Criteria:

1. Currently receiving or have within the past 2 month received radio- and/or chemotherapy
2. Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.
3. Are pregnant or breastfeeding
4. Having dermatological problems in the peristomal- or abdominal area (assessed by investigating scientist)
5. Participating in other interventional clinical investigations or have previously participated in this evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2017-02-09 (Actual)

PRIMARY OUTCOMES:
Trans epidermal water loss | 6 hours
  The condition of the skin is measure by trans epidermal water loss after removing the adhesive strip.

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Nielsen, M. Sci, Principal Investigator — Head of preclinical department
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

IPD SHARING:
Plan to Share IPD: No